CLINICAL TRIAL: NCT04362995
Title: SJTRC-St. Jude Tracking of Viral and Host Factors Associated With COVID-19: A Prospective Adaptive Cohort Study
Brief Title: St. Jude Tracking of Viral and Host Factors Associated With COVID-19
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Georgia (Other); University of Wisconsin, Madison (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: SJTRC; NIH1P01AI165077-01 (Other: Sub-award from University of Wisconsin, Madison); 75N93019C00052 (Other: Sub-award from University of Georgia); 5R01AI136514-05 (NIH); 75N93021C00016 (Other Grant/Funding Number: Contract Number - CEIRR NIAID program)
Record Dates: First submitted 2020-04-22; First posted 2020-04-27 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Coronavirus Infection; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, and nasal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SARS-CoV-2 Infection: St. Jude Children's Research Hospital employees with SARS-CoV-2 infection
- Controls: St. Jude Children's Research Hospital employees uninfected with SARS-CoV-2 infection
- Long Term Follow Up (LTFU): Subset of participants who participated in the original SJTRC study and agree to continue in LTFU

SUMMARY:
This is a prospective adaptive cohort study of St. Jude employees to determine the rate of SARS-CoV-2 infections that are asymptomatic and to evaluate immunological responses to SARS-CoV-2 infection.

Primary Objectives

* To estimate the proportion of asymptomatic infection with SARS-CoV-2 infection in a population of SARS-CoV-2-naïve adult St. Jude employees
* To comprehensively map CD4 and CD8 T cell epitopes and response magnitudes to SARS-CoV-2 infection in a population of SARS-CoV-2-naïve adult St. Jude employees who acquire SARS-CoV-2 infection
* To measure changes in the CD4 and CD8 response magnitude and function to SARS-CoV-2 infection and/or vaccination in a population of St. Jude employees for up to 48 months after infection and/or vaccination.

Secondary Objectives

* To establish seroprevalence of SARS-CoV-2-specific antibodies at baseline, and identify the rate of seroconversion to SARS-CoV-2 in a population of presumably naïve adult St. Jude employees
* To identify features of T cell responses at baseline and during SARS-CoV-2 infection that are associated with protection against symptomatic or severe COVID-19 disease in a population of adult St. Jude employees
* To identify risk factors for long-term protection against COVID-19 in a population of adult St. Jude employees
* To evaluate changes in antibody responses to SARS-CoV-2 in a population of St. Jude employees for up to 48 months after SARS-CoV-2 infection and/or vaccination.
* To evaluate the saliva antibody and cytokine response to SARS-CoV-2 infection and/or vaccination and identify characteristics that predict protection from subsequent SARS-CoV-2 infection among a population of St. Jude employees followed for up to 48 months after SARS-CoV-2 infection and/or vaccination.
* To measure changes in saliva antibody responses to SARS-CoV-2 for up to 48 months after SARS-CoV-2 infection and/or vaccination.

Exploratory Objectives

* To establish additional immunological features including host immune or receptor polymorphisms associated with response to SARS-CoV-2 infection
* To explore SARS-CoV-2 diversity and specific features in a circumscribed population
* To describe the presence, characteristics, and proportion of short-term re-infection
* To determine if an association between SARS-CoV-2 viral load in nasal swab specimens and COVID-19 symptoms can be identified in a population of adult St. Jude employees who acquire SARS-CoV-2
* To explore the laboratory and clinical response to SARS-CoV-2 vaccine in a population of adult St. Jude employees with and without a history of SARS-CoV-2 infection

DETAILED DESCRIPTION:
Naive individuals will contribute a baseline blood sample at enrollment. Subsequent routine blood draws will occur to determine the proportion of participants who have asymptomatically seroconverted; the timing of these blood draws and proportion of participants required will be determined by the rate of documented SARS-CoV-2 infection in the cohort according to an adaptive study design. Participants will be tracked for SARS-CoV-2 specific antibodies and CD4, and CD8 T cell responses throughout the period and especially during the early stages after clearance of infection and subsequently to determine the quality and duration of memory responses.

In addition to blood samples, participants will intermittently provide nasal swabs for detection of SARS-CoV-2; this will occur either through a comprehensive proactive employee screening program, or specifically for the purposes of the research study if participants are required to attend campus but are not currently eligible for employee screening. These will determine duration and characteristics of viral shedding and identify reinfection. Seroprevalence estimates and asymptomatic conversion will also be determined.

Individuals with a diagnosis of COVID-19 infection will have two additional blood draws in the acute and convalescent phase to identify acute and late immune responses. These responses will be compared to the essential baseline sample data to characterize the generation of de novo and cross-reactive recall responses.

For those participants receiving vaccination, blood draws will be taken after COVID vaccine (3-8 weeks after completion of 1 or 2 dose course) and at completion of study.

At enrollment, subjects will complete a baseline online personal health and demographic questionnaire, and then monthly brief online health update questionnaires. Throughout the study period, subjects will complete a brief online symptom survey every 2 weeks.

Participants in the original SJTRC study will be asked to reconsent to complete a one-time questionnaire regarding their COVID-19 experience specifically during the time since they went off study. Once this questionnaire is complete, they will be taken off study and receive no further questionnaires related to the original study.

A subset of participants will be invited to re-enroll in a long-term follow-up phase to evaluate long-term immunity and protection against COVID-19 following infection and vaccination. Participants will provide blood samples every 6 months. They will also be invited to provide additional acute and convalescent samples (blood and saliva), if diagnosed with acute COVID-19 during this period. Participants will continue to complete regular questionnaires, but the frequency will decrease to 6 monthly (health questionnaires) and as needed (COVID-19 diagnosis or vaccination).

ELIGIBILITY:
Inclusion Criteria:

1. Adult St. Jude employees (Age ≥ 18 years of age) who are presumed to be SARS- CoV-2 naive, or have a recent diagnosis of COVID-19, and volunteer to participate.
2. Willing to undergo blood draws on up to 5 occasions during the study.
3. Receiving approximately twice-weekly SARS-CoV-2 screening by Occupational Health, or willing to provide up to twice weekly nasal self-swabs if attending campus.
4. Have access to a personal smartphone that is able to receive and respond to text messages for data collection.
5. Has ready access to the internet to log personal study information into the REDCap database.
6. Self-identified as able to speak and read English well enough to understand the consent process and survey forms, and to report symptoms.

Inclusion Criteria for LTFU arm:

1. Adult St. Jude employees (age ≥ 18 years of age) who participated in the original SJTRC study.
2. Willing to undergo blood draws on up to five occasions during the LTFU arm. Willing to provide saliva samples at acute and convalescent episodes.
3. Have access to a personal smartphone that is able to receive and respond to text messages for data collection.
4. Have ready access to the internet to log personal study information into the REDCap database.
5. Self-identified as able to speak and read English well enough to understand the consent process and questionnaires, and to report symptoms.

Exclusion Criteria:

1. Employees who are first-degree relatives of, or directly or indirectly report up to, the PI or any of the clinical study investigators who will have access to participant identities.
2. Employees who cannot complete the informed consent process.

Exclusion Criteria for LTFU arm:

1. Employees who did not participate in the original SJTRC study.
2. Employees who cannot complete the informed consent process.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: St. Jude employees who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1316 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Proportion of asymptomatic subjects | 1 year from enrollment
  The proportion of participants who test positive for SARS-CoV-2 infection but remain asymptomatic.
Positive CD4 and CD8 cell epitope positive response | at enrollment, 3 months, 6 months, 9 months and 1 year
  A list of CD4 and CD8 cell epitopes with a magnitude change from baseline that is at least twice the standard deviation of the baseline.
Positive CD4 and CD8 cell epitope positive response | up to 48 months of additional observation in participants who have had COVID-19 or vaccination
  A list of CD4 and CD8 cell epitopes with a magnitude change from baseline that is at least twice the standard deviation of the baseline.

SECONDARY OUTCOMES:
Proportion of seroprevalence | Baseline, 3 months, 6 months, 9 months and 1 year
  The proportion of participants at each time point who have detectable antibodies that recognize SARS-COV-2.
T-cell response | Baseline, 3 months, 6 months, 9months, 1 year and 6 monthly for an additional 48 months in participants included in the long-term follow-up arm
  For CD8s, T cell responses will be categorized as cytolytic, cytokine producing, or exhausted. For CD4s they will be grouped as Th1, Th2, Tfh, or Th17. Percentages of cells in each category will be summarized at baseline and during SARS-CoV-2 infection.
Protective antibody responses against SARS-CoV-2 at last follow-up sample | up to 48 months of additional observation in participants who have had COVID-19 or vaccination
  For participants who have enrolled in the long-term follow-up arm of the study, associations between persistent protective antibody responses and clinical and laboratory characteristics will be evaluated by paired tests and regression models.
Change in antibody responses to SARS-CoV-2 | up to 48 months of additional observation in participants who have had COVID-19 or vaccination
  For participants who have enrolled in the long-term follow-up arm of the study, changes in antibody levels from baseline in paired samples.
Saliva antibody and cytokine responses to SARS-CoV-2 | up to 48 months of additional observation in participants who have had COVID-19 or vaccination
  For participants who have enrolled in the long-term follow-up arm of the study, changes in saliva antibody and cytokine levels from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Paul G. Thomas, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Schultz-Cherry S, McGargill MA, Thomas PG, Estepp JH, Gaur AH, Allen EK, Allison KJ, Tang L, Webby RJ, Cherry SD, Lin CY, Fabrizio T, Tuomanen EI, Wolf J; SJTRC Investigative Team. Cross-reactive Antibody Response to mRNA SARS-CoV-2 Vaccine After Recent COVID-19-Specific Monoclonal Antibody Therapy. Open Forum Infect Dis. 2021 Aug 10;8(9):ofab420. doi: 10.1093/ofid/ofab420. eCollection 2021 Sep. PMID 34557558
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols